CLINICAL TRIAL: NCT07401238
Title: Piezo-assisted Expansion of Narrow Ridges for Implant-supported Treatment of Intercalated Mono-edentulism: A Case Series Study
Brief Title: Piezo-assisted Expansion of Narrow Ridges
Acronym: PRIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Trieste (Other)
Collaborators: International Piezosurgery Academy (Other)
Responsible Party: Principal Investigator, prof. Roberto Di Lenarda, prof, University of Trieste
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 55/2016
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Bone Atrophy, Alveolar
Keywords: implant; alveolar ridge expansion; graft
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: case series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- narrow ridge (Experimental): width comprised between 3 and 5 mm
  Interventions: Procedure: Alveolar Ridge Reconstruction

INTERVENTIONS:
Procedure: Alveolar Ridge Reconstruction — wedge shaped xenograft inserted in splitted alveolar crest
  Other Names: split crest

SUMMARY:
the goal of the study was the evaluation of the clinical and histological performance of delayed inserted implants in augmented sites with a shaped solid graft inserted in an originally narrow alveolar edentulous ridge.

DETAILED DESCRIPTION:
Purpose To assess the efficacy of a two-stage piezo-assisted split crest technique and delayed implant insertion. Computed tomography, radiological, clinical, and histologic evaluation.

Research design Multicenter case-series

Sample size 20 patients People involved in the protocol At least 25 enrolled patients (5 per center) counting drop-outs

Inclusion criteria

1. Patients with single mandibular or maxillary intercalated edentulism (1 implant) who require implant rehabilitation with conventional loading
2. The edentulous site width should be comprised between 3 and 5mm for the first 3mm of height
3. Presence of visible spongious bone in CBCT cross-sections
4. The edentulous site must present at least 4mm wide band of keratinized tissue
5. Plaque index < 20%, Bleeding index < 25%
6. Medical condition of the enrolled patients should be within ASA 2 score
7. Only no smokers, light smokers (< 10 per day) or electronic smokers will be accepted

Exclusion criteria

1. Head and neck RT in the previous 5 years
2. Previous or actual antiresorptive therapy
3. Chronic corticosteroid therapy
4. Pregnancy or breastfeeding
5. Active periodontal disease
6. Abuse of alcohol or drugs
7. Incapability of understanding the purposes of the study (e.g. mental deficit)

Evaluation criteria

1. Presurgical evaluation with low-dose CBCT scan of the edentulous site
2. Intraoperative evaluation of crestal bone width before and after crest-splitting
3. Presurgical (second stage) CBCT scan before implant placement
4. Histologic and histomorphometric evaluation of bone samples harvested during implant site preparation
5. Implant stability: IT (insertion torque) and ISQ (implant stability quotient)
6. Marginal bone loss assessed with intraoral radiographies at implant placement, at prosthetic loading, after 6 months, 1, 2 and 3 years after loading

Data analysis The continuous variables will be expressed with average, median and standard deviation. Categorical variables will be expressed in numbers and percentages. There are parametrical and non parametrical statistical tests.

PREFACE

Ridge expansion (split crest or crest-splitting) is used to widen narrow ridges with adequate height for implant placement. This human case series presents radiologic, clinical and histologic results of delayed implant placement after ridge expansion and grafting of single implant sites with piezoelectric bone surgery. Bone expansion in oral surgery consists of expanding the atrophic bone crest to obtain sufficient bone width for proper dental implant placement. To achieve this result, different regenerative surgical techniques have been developed: conventional onlay/inlay grafts, interpositional sandwich osteotomies, guided bone regeneration with semipermeable membranes and alveolar distraction osteogenesis. All these procedures can be used for alveolar ridge augmentation with autologous or homologous bone grafts, xenografts, or synthetic bone substitutes to allow implant placement in one or two surgical steps. Even if the survival rate of implants inserted in expanded crests was reported to be almost 100% after 5 years of loading, several protocols have been proposed (one stage, two stage, with or without graft) together with different surgical devices (manual osteotomy, surgical burs, piezoelectric devices). One of the most critical aspects of the technique is the bone vascularization after expansion, together with the vestibular plate integrity and the long term peri-implant bone stability.

STUDY PURPOSES The primary purpose of this study is the evaluation of the effects on implant survival and prevalence of complications of a two-stage ridge expansion technique with piezoelectric dedicated tips, xenograft positioning and surgical re-entry after four months for implant placement.

MATERIALS Diagnostic and surgical instruments kit CBCT scans will be performed using last generation devices with low-dose protocol. Acteon Cube by Acteon-Satelec will be used as piezoelectric device. "Crest-splitting" tips will be used for ridge expansion, according to the manufacturer's instructions. A commercially available wedge shaped xenograft (cancellous equine collagenated bone; V-Block, Tecnoss, Italy) will be inserted between the splitted corticals as a space maintainer. A commercially available cross-linked bovine collagen membrane (Evolution, Tecnoss, Italy) will be used to cover the surgical site. 6/0 monofilament suture will be used for wound closure. After 5 months of healing, a stainless steel trephine bur mounted on an implant handpiece (4 mm external diameter, 3 mm internal diameter) will be used for implant site preparation. Bone samples harvested to prepare implant site will be stored immediately in 4% buffered formalin. A commercially available tapered implant of 3.5 mm diameter with conical connection will be positioned in the prepared site (M2, Zeros, South Korea). After 3 months of submerged healing, implants will be uncovered and restored with screwed ceramic single crowns.

EU marking All the products used in this study are marked EU and available for sale. Traceability On each package there is a label that can be attached to each patient schedule for a complete traceability of the product.

STUDY DESIGN

* The design is case series
* All the patients have to sign the authorization to use and process their own personal details.
* All biomaterials used in this study are available on the market
* All the products used are EU marked
* There must be treated at least 25 patients
* The participants must be selected in respect of the inclusion and exclusion criteria
* The experimenter must inform all the participants about the treatment of this study and receive an informed consent by them.

NUMBER OF PARTICIPANTS Sample size The minimal number of the participants of this study is 20; expecting dropouts of 1 patient per center will give a total of 25 patients. The sample must be enrolled in 24 months.

Number of Centers Five centers

Duration of the study The study can start on May 2020. The sample must be enrolled within 12 months. The follow-up time will be 3 years after loading of the implants; the total time estimated to complete the study is 5 years.

Follow-up timing Follow-up Control code Time Pre-surgical CBCT evaluation C0 Time 0 (T0) Intra-operative evaluation (stage1) C1 Time 1 (T1) Post-surgical CBCT evaluation (stage2) C2 Time 2 (T2) after 5 months from T1 Intra-operative evaluation (stage2) C3 Time 3 (T3) after 5 months from T1 Loading phase C4 Time 4 (T4) after 3 months from T3 6 months post loading C5 Time 5 (T5) 12 months post loading C6 Time 6 (T6) 24 months post loading C7 Time 7 (T7) 36 months post loading C8 Time 8 (T8)

Methods SELECTION OF PATIENTS Inclusion criteria

1. Patients with single mandibular or maxillary intercalated edentulism (1 implant) who require implant rehabilitation with conventional loading
2. The edentulous site width should be comprised between 3 and 5mm for the first 3mm of height
3. Presence of visible spongious bone in CBCT cross-sections
4. The edentulous site must present at least 4mm wide band of keratinized tissue
5. Plaque index < 20%, Bleeding index < 25%
6. Medical condition of the enrolled patients should be within ASA 2 score
7. Only no smokers, light smokers (< 10 per day) or electronic smokers will be accepted

Exclusion criteria

1. Head and neck RT in the previous 5 years
2. Previous or actual antiresorptive therapy
3. Chronic corticosteroid therapy
4. Active periodontal disease
5. Pregnancy or breastfeeding
6. Abuse of alcohol or drugs
7. Incapability of understanding the purposes of the study (e.g. mental deficit)

   Information for the patients The patients will be informed about the treatment, the benefits and the possible risks. The patients will be told that the clinical data collected during the pre- and post- implant surgery will be used for a clinical study and should authorize the use and processing of these data. The use of these details will strictly respect the anonymity, and will be always strictly confidential and exclusive for the purpose of the study. A copy of the informed consent form is kept by the experimenter, and another copy is for the patient.

   Evaluation The data contained in the "Case Report Form" report the pre-surgery analysis and the information collected during the peri-operatory period in each enrolled patient.

   Basic data

   These are the collected and documented data:
   * Date of the control
   * Identification number of the patient preceded by the univocal letters of the center "xX" with a progressive number. Center codes will be: TS (University of Trieste), GO (Claudio Stacchi), HD (Teresa Lombardi), SM (Simone Verardi).

   Details for test group only A) Pre-operating data

   • Obtaining informed consent
   * Obtaining authorization to use and process personal details
   * Assignment of the patient code in the CRF form

   General data

   • Remote medical history
   * Edentulism
   * Pathologies (if present)
   * Pharmacological therapy

   Radiological data

   • Cone beam CT in DICOM format, mandatory for the inclusion of the patient (coronal 3mm of the crest comprised between and 5mm of width).

   Clinical evaluation:
   * Plaque index
   * Bleeding index
   * PSR (periodontal screening and recording)

   B) Intra-operative data

   • Systemic and local prophylaxis (antibiotics, disinfectants, anti-inflammatories, etc.). An antibiotic coverage therapy for 6 days from one hour after the procedure with Augmentin 1gr (2 tablets/day) or Clindamycin 600 mg (1 tablet/day) is mandatory.

   • Anesthesia technique

   • Flap design: full thickness

   • Number of piezo tips used to gain the final expansion (all, all but the last, etc.)

   • Implant insertion after bone harvesting

   • Registration of IT and ISQ at T3

   • Healing abutment positioning (if IT>30, ISQ >65)

   • Intra-operative complications (for instance: cortical perforation, evident fixture mobility during the placement, neurological complications, etc.)
   * Periapical radiograph at the moment of implant placement using a Rinn holder and a silicon individual stent (to be delivered to the patients for every examination)
   * Measuring of ISQ at T4 (impression phase) and radiograph
   * Radiographic evaluation during follow up timepoints
   * Clinical evaluation during follow up timepoints (6-sites peri-implant probing, IP and BoP).
   * Exemplificative iconographic evaluation.

   C) Post-operative data • Clinical evaluation These information are written in the CRF

   Complications

   • Type of complication

   • Start, end and course

   • Seriousness
   * Therapy
   * Relationship with the fixture or the surgical instrumentation

   Case closing • Reason of the closing
   * Date of the last control
   * Date of the closing

   Statistic processing The demographic variables and the clinical continuous data are processed with medium and median value and with standard deviations. Categorical variables are processed with frequency charts and percentages. Data normality will be assessed by using Kolmogorov-Smirnov test and equality of variances by using Levene test. Parametric and non-parametric statistic tests for repeated measures will be used.

   Adverse events and reactions The experimenter has the responsibility to report immediately all the adverse events or reactions related to the products during the study period. An adverse event or reaction is considered serious if it brings a permanent damage to the patient or if it makes a second operation necessary. All the adverse events or reactions should be communicated writhing within a short time through letters, faxes or e-mails to the appropriate authority or to the coordinator experimenter

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with single mandibular or maxillary intercalated edentulism (1 implant) who require implant rehabilitation with conventional loading 2. The edentulous site width should be comprised between 3 and 5mm for the first 3mm of height 3. Presence of visible spongious bone in CBCT cross-sections 4. The edentulous site must present at least 4mm wide band of keratinized tissue 5. Plaque index < 20%, Bleeding index < 25% 6. Medical condition of the enrolled patients should be within ASA 2 score 7. Only no smokers, light smokers (< 10 per day) or electronic smokers will be accepted

Exclusion Criteria:

* 1. Head and neck RT in the previous 5 years 2. Previous or actual antiresorptive therapy 3. Chronic corticosteroid therapy 4. Active periodontal disease 5. Pregnancy or breastfeeding 6. Abuse of alcohol or drugs 7. Incapability of understanding the purposes of the study (e.g. mental deficit)

Max Age: 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2026-02-03 (Actual); Study Completion 2026-02-03 (Actual)

PRIMARY OUTCOMES:
postoperative surgical width | 5 months
  radiologically measured alveolar expansion

SECONDARY OUTCOMES:
new bone formation | 5 months later than surgery
  histomorphometric analysis

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li X, Xu P, Xu X, Liu S. The application of a delayed expansion technique for horizontal alveolar ridge augmentation in dental implantation. Int J Oral Maxillofac Surg. 2017 Nov;46(11):1451-1457. doi: 10.1016/j.ijom.2017.05.025. Epub 2017 Jun 26. PMID 28663017